CLINICAL TRIAL: NCT02190903
Title: A Randomized Controlled Trial To Assess Risk of Delirium in Older Adults Undergoing Hip Fracture Surgery With Spinal or General Anesthesia
Brief Title: A Trial To Assess Risk of Delirium in Older Adults Undergoing Hip Fracture Surgery With Spinal or General Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Mark Neuman, Assistant Professor of Anesthesiology and Critical Care, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 818017
Record Dates: First submitted 2014-06-30; First posted 2014-07-15 (Estimated); Results first posted 2018-07-30 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Postoperative Complications; Hip Fracture; Delirium
Keywords: delirium; hip fracture; general anesthesia; spinal anesthesia; postoperative complications
MeSH Terms: conditions — Postoperative Complications; Hip Fractures; Delirium | interventions — Amino Acid Motifs; Anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- General endotracheal anesthesia (Active Comparator): Standard care general endotracheal anesthesia
  Interventions: Other: General endotracheal anesthesia
- Regional (spinal) anesthesia (Active Comparator): Standard care spinal anesthesia
  Interventions: Other: Regional (spinal) Anesthesia

INTERVENTIONS:
Other: General endotracheal anesthesia — General Anesthesia
  Patients randomized to receive general anesthesia induction of anesthesia with intravenous lidocaine, propofol, fentanyl citrate and vecuronium or cisatracurium, following dosing guidelines defined by protocol. Following tracheal intubation, anesthesia will be maintained with sevoflurane in oxygen and air as defined by protocol. End-tidal gas monitoring (for carbon dioxide and sevoflurane) and maintenance, monitoring, and reversal of neuromuscular blockade will be as per HUP and PPMC routine. Immediate postoperative analgesia will be via IV dilaudid dosed intraoperatively as defined by protocol.
  Arms: General endotracheal anesthesia
Other: Regional (spinal) Anesthesia — Patients randomized to receive spinal anesthesia will undergo spinal blockade using standard techniques and medications dosed as per protocol, and will include hyperbaric bupivicaine or tetracaine, fentanyl citrate, and epinephrine; algorithms for management of spinal-related hypotension will be defined by protocol. Intraoperative sedation will be achieved via continuous intravenous propofol infusion; supplemental oxygen will be provided by nasal cannula or facemask as needed.
  Arms: Regional (spinal) anesthesia

SUMMARY:
This pilot project will address the gaps in knowledge regarding the effect of anesthetic technique on the risk of delirium through an adequately-powered trial employing standardized regimens for treatment and outcome assessment to test the hypothesis that use of spinal versus general anesthesia decreases the risk of delirium after hip fracture surgery.

DETAILED DESCRIPTION:
Objectives Overall objectives Overall Objectives Specific Aims

1. To compare the effect of spinal versus general anesthesia on rates of postoperative delirium after hip fracture surgery. We hypothesize that rates of delirium after hip fracture surgery will be lower among patients receiving spinal versus general anesthesia.
2. To develop, field-test, and conduct a qualitative evaluation of protocols and procedures for a planned multicenter trial to test the association of anesthesia technique with survival and recovery of function in activities of daily living ambulatory ability at six months after hip fracture.

Primary outcome variable(s) The primary outcome variable is the rate of delirium after hip fracture surgery.

Background Delirium, or a disturbance of consciousness and a change in cognition that develop over a short period of time, (1) complicates 2.6 million hospitalizations among U.S. adults aged 65 or older each year. (2,3) Patients who experience delirium during hospitalization face increased risks morbidity, mortality, and functional disability. (4) Each year, delirium accounts for $6.9 billion in Medicare hospital expenditures. (5) Delirium occurs in 35% to 65% of the 320,000 older U.S. adults hospitalized for hip fracture each year. (6) While adverse survival and functional outcomes are common after hip fracture, (7) a single episode of delirium doubles the odds of both new functional dependence and new ambulatory disability at six months after fracture, and triples the odds of death or new nursing home placement. (8) Compared to general endotracheal anesthesia, spinal anesthesia may decrease the incidence of postoperative delirium after hip fracture surgery. Small randomized trials of anesthesia type for hip fracture have suggested a 50% lower risk of acute confusion after hip fracture surgery with spinal anesthesia, (9) but the heterogeneity of outcome definitions and measurement strategies employed by past trials, along with their use of historical anesthesia practices limit their applicability to current practice.

As a result of these limitations, clinical equipoise continues to exist regarding the optimal anesthetic technique for hip fracture care. Compared to general anesthesia, spinal anesthesia may offer potential benefits not limited to decreased delirium. These may include decreased intraoperative blood loss, and decreased risks of postoperative thromboembolic events, respiratory infections and malignant hyperthermia. At the same time, spinal anesthesia may be associated with greater hypotension than general anesthesia, and may carry small risks of bleeding and infection at the site of the spinal injection and discomfort during block placement. Relative to spinal anesthesia, general anesthesia may offer benefits of hemodynamic stability. At present, while spinal anesthesia has been demonstrated in a retrospective observational study to be associated with lower in-hospital mortality after hip fracture (10), a meta-analysis of randomized trials was inconclusive with regard to mortality differences. (9) Reflecting this state of clinical equipoise patterns of anesthesia care differ widely by country and by provider, reflecting a large role of provider practice style in determining anesthesia care for hip fracture. For example, in a recent survey of UK anesthesiologists, 76% indicated that they routinely performed hip fracture surgeries with spinal anesthesia (11). In contrast, recent U.S. data suggest that approximately 80% of hip fracture surgeries are performed with general anesthesia, with wide variability in practice across hospitals.(10) While these variations may in part reflect differences in patient preferences, the current state of knowledge regarding the risks and benefits of differing types of anesthesia is inadequate to support appropriately informed medical decision-making by either patients or health care providers. The UKs national institute for Health and Care Excellence (NICE) strongly recommend further clinical trials to provide additional information regarding the clinical and cost effectiveness of differing anesthesia types for hip fracture, stating that they were unable to identify any recent randomised controlled trialsthat fully address this question and that the [available] evidence is old and does not reflect current practice.

Study Design Phase II

Design This is a randomized, controlled trial of spinal versus general anesthesia to test the effect of anesthesia type on rates of postoperative delirium after hip fracture surgery.

Study duration It is expected that this study will begin enrollment in June 2013. The enrollment of all subjects is projected to be completed in May 2014 with data analysis to follow. The study will hope to be completed by June 2015.

The length of participation for each subject will be about 5 days.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is aged 18 and older.
2. Subject is scheduled to undergo surgical treatment of an acute femoral neck or pertrochanteric hip fracture.
3. Subject can speak English
4. Subject has ability to sign informed consent

Exclusion Criteria:

1. Subject has a pathological or periprosthetic fracture.
2. Subject has concurrent conditions anticipated at the time of admission to require surgical treatment (e.g. multiple trauma, acute cholecystitis).
3. Subject has severe cognitive impairment, as evidenced by a Montreal Cognitive Assessment Score (MOCA) of 15 or less.
4. Subject has clinical findings of delirium prior to surgery, as evidenced by a positive Confusion Assessment Method (CAM) evaluation;
5. Subject has contraindications to spinal anesthesia or volatile general anesthetics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-10; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark D Neuman, Principal Investigator — University of Pennsylvania
Locations (1):
- Hosptial of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] American Psychiatric Association. Delirium, Dementia, and Amnestic and Other Cognitive Disorders. In: Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (Text Revision). Washington, D.C.: American Psychiatric Association; 2000.
- [Background] Russo CA, Elixhauser A. Hospitalizations in the Elderly Population, 2003. 2006 May. In: Healthcare Cost and Utilization Project (HCUP) Statistical Briefs [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2006 Feb-. Statistical Brief #6. Available from http://www.ncbi.nlm.nih.gov/books/NBK63501/ PMID 21938846
- [Background] Fong TG, Tulebaev SR, Inouye SK. Delirium in elderly adults: diagnosis, prevention and treatment. Nat Rev Neurol. 2009 Apr;5(4):210-20. doi: 10.1038/nrneurol.2009.24. PMID 19347026
- [Background] Inouye SK, Rushing JT, Foreman MD, Palmer RM, Pompei P. Does delirium contribute to poor hospital outcomes? A three-site epidemiologic study. J Gen Intern Med. 1998 Apr;13(4):234-42. doi: 10.1046/j.1525-1497.1998.00073.x. PMID 9565386
- [Background] Inouye SK. Delirium in older persons. N Engl J Med. 2006 Mar 16;354(11):1157-65. doi: 10.1056/NEJMra052321. No abstract available. PMID 16540616
- [Background] Blackman DK, Kamimoto LA, Smith SM. Overview: surveillance for selected public health indicators affecting older adults--United States. MMWR CDC Surveill Summ. 1999 Dec 17;48(8):1-6. PMID 10634268
- [Background] Hung WW, Egol KA, Zuckerman JD, Siu AL. Hip fracture management: tailoring care for the older patient. JAMA. 2012 May 23;307(20):2185-94. doi: 10.1001/jama.2012.4842. PMID 22618926
- [Background] Marcantonio ER, Flacker JM, Michaels M, Resnick NM. Delirium is independently associated with poor functional recovery after hip fracture. J Am Geriatr Soc. 2000 Jun;48(6):618-24. doi: 10.1111/j.1532-5415.2000.tb04718.x. PMID 10855596
- [Background] Parker MJ, Handoll HH, Griffiths R. Anaesthesia for hip fracture surgery in adults. Cochrane Database Syst Rev. 2004 Oct 18;(4):CD000521. doi: 10.1002/14651858.CD000521.pub2. PMID 15494999
- [Background] Neuman MD, Silber JH, Elkassabany NM, Ludwig JM, Fleisher LA. Comparative effectiveness of regional versus general anesthesia for hip fracture surgery in adults. Anesthesiology. 2012 Jul;117(1):72-92. doi: 10.1097/ALN.0b013e3182545e7c. PMID 22713634
- [Background] Sandby-Thomas M, Sullivan G, Hall JE. A national survey into the peri-operative anaesthetic management of patients presenting for surgical correction of a fractured neck of femur. Anaesthesia. 2008 Mar;63(3):250-8. doi: 10.1111/j.1365-2044.2007.05328.x. PMID 18289230
- [Background] National Clinical Guideline Centre (UK). The Management of Hip Fracture in Adults [Internet]. London: Royal College of Physicians (UK); 2011. Available from http://www.ncbi.nlm.nih.gov/books/NBK83014/ PMID 22420011
- [Background] Sieber FE, Zakriya KJ, Gottschalk A, Blute MR, Lee HB, Rosenberg PB, Mears SC. Sedation depth during spinal anesthesia and the development of postoperative delirium in elderly patients undergoing hip fracture repair. Mayo Clin Proc. 2010 Jan;85(1):18-26. doi: 10.4065/mcp.2009.0469. PMID 20042557
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Inouye SK, van Dyck CH, Alessi CA, Balkin S, Siegal AP, Horwitz RI. Clarifying confusion: the confusion assessment method. A new method for detection of delirium. Ann Intern Med. 1990 Dec 15;113(12):941-8. doi: 10.7326/0003-4819-113-12-941. PMID 2240918
- [Background] Kernan WN, Viscoli CM, Makuch RW, Brass LM, Horwitz RI. Stratified randomization for clinical trials. J Clin Epidemiol. 1999 Jan;52(1):19-26. doi: 10.1016/s0895-4356(98)00138-3. PMID 9973070
- [Background] Simon R. Restricted randomization designs in clinical trials. Biometrics. 1979 Jun;35(2):503-12. PMID 486683
- [Background] Sessler CN, Gosnell MS, Grap MJ, Brophy GM, O'Neal PV, Keane KA, Tesoro EP, Elswick RK. The Richmond Agitation-Sedation Scale: validity and reliability in adult intensive care unit patients. Am J Respir Crit Care Med. 2002 Nov 15;166(10):1338-44. doi: 10.1164/rccm.2107138. PMID 12421743
- [Background] KATZ S, FORD AB, MOSKOWITZ RW, JACKSON BA, JAFFE MW. STUDIES OF ILLNESS IN THE AGED. THE INDEX OF ADL: A STANDARDIZED MEASURE OF BIOLOGICAL AND PSYCHOSOCIAL FUNCTION. JAMA. 1963 Sep 21;185:914-9. doi: 10.1001/jama.1963.03060120024016. No abstract available. PMID 14044222
- [Background] Inouye SK, Viscoli CM, Horwitz RI, Hurst LD, Tinetti ME. A predictive model for delirium in hospitalized elderly medical patients based on admission characteristics. Ann Intern Med. 1993 Sep 15;119(6):474-81. doi: 10.7326/0003-4819-119-6-199309150-00005. PMID 8357112
- [Background] Kahan BC, Morris TP. Improper analysis of trials randomised using stratified blocks or minimisation. Stat Med. 2012 Feb 20;31(4):328-40. doi: 10.1002/sim.4431. Epub 2011 Dec 4. PMID 22139891

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 15 patients provided informed consent for participation; 3 were withdrawn from the study prior to randomization. 2 of these patients were withdrawn due to ineligibility; 1 was withdrawn due to other reasons.
Groups:
- General Endotracheal Anesthesia: Standard care general endotracheal anesthesia
  General endotracheal anesthesia: General Anesthesia
  Patients randomized to receive general anesthesia induction of anesthesia with intravenous lidocaine, propofol, fentanyl citrate and vecuronium or cisatracurium, following dosing guidelines defined by protocol. Following tracheal intubation, anesthesia will be maintained with sevoflurane in oxygen and air as defined by protocol. End-tidal gas monitoring (for carbon dioxide and sevoflurane) and maintenance, monitoring, and reversal of neuromuscular blockade will be as per HUP and PPMC routine. Immediate postoperative analgesia will be via IV dilaudid dosed intraoperatively as defined by protocol.
- Regional (Spinal) Anesthesia: Standard care spinal anesthesia
  Regional (spinal) Anesthesia: Patients randomized to receive spinal anesthesia will undergo spinal blockade using standard techniques and medications dosed as per protocol, and will include hyperbaric bupivicaine or tetracaine, fentanyl citrate, and epinephrine; algorithms for management of spinal-related hypotension will be defined by protocol. Intraoperative sedation will be achieved via continuous intravenous propofol infusion; supplemental oxygen will be provided by nasal cannula or facemask as needed. Propofol dose will be titrated to achieve light to moderate sedation, defined as a Richmond Agitation/Sedation Scale (RASS) score of -1 to -318. In the event of block failure induction and maintenance of general endotracheal anesthesia will occur via the procedures outlined above. For all patients, post-operative pain management will be via hydromorphone PCA or PRN hydromorphone bolus, followed by oral oxycodone and acetaminophen.
Period: Overall Study
Arm/Group | General Endotracheal Anesthesia | Regional (Spinal) Anesthesia
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | General Endotracheal Anesthesia | Regional (Spinal) Anesthesia | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 62.7 [57 to 88] | 80.5 [62 to 92] | 71.5 [62 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 5 | 4 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Postoperative Delirium After Hip Fracture Surgery
Description: Delirium will be assessed by the Confusion Assessment Method Instrument (CAM), a validated method of assessing delirium based on the presence of both (1) an acute onset of signs and symptoms with a fluctuating course AND (2) inattention; PLUS (3) disorganized thinking OR (4) an altered level of consciousness.
Time Frame: Up to 5 days post hip fracture surgery
Measure: Count of Participants; unit: Participants
Arm/Group | General Endotracheal Anesthesia | Regional (Spinal) Anesthesia
Number analyzed (Participants) | 6 | 6
Participants | 2 | 0

ADVERSE EVENTS:
Arm/Group | General Endotracheal Anesthesia | Regional (Spinal) Anesthesia
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | General Endotracheal Anesthesia (N=6) | Regional (Spinal) Anesthesia (N=6)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
This was a limited pilot study conducted to assess the feasibility of a larger randomized trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes